CLINICAL TRIAL: NCT07115680
Title: Countries Where the Main Authors and Their Collaborators of Recently Published Clinical Pharmacology Studies Worked
Brief Title: Where Did the Authors Work When They Conducted Their Clinical Pharmacology Studies?
Status: Completed | Type: Observational
Sponsor: Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz (Other)
Responsible Party: Sponsor
Other Study IDs: IIS-FJD-RDR-2025-001
Record Dates: First submitted 2025-08-04; First posted 2025-08-11 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Scientific Collaboration in Clinical Pharmacology
Keywords: Clinical pharmacology, studies on humans, recently published

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single-country studies: Multinational studies
  Interventions: Other: human participants, data or material

INTERVENTIONS:
Other: human participants, data or material — Articles on human participants, data, or material published in top (as per JCR IF) clinical pharmacology journals linked to professional societies

SUMMARY:
It is unknown in which countries the clinical pharmacology studies published in leading specialized journals were conducted. The hypothesis is that studies in this specialty tend to be conducted and published by authors from a single country. This analysis aims to describe the number of collaborators and the countries in which they worked, using the Nature Index concept of "share."

DETAILED DESCRIPTION:
Original articles (full reports, short communications, research letters) on human participants, data, or material published in the seven top (as per Journal Citations Report 2024 Impact Factor) clinical pharmacology hybrid journals linked to clinical pharmacology professional societies will be included. Articles of interest to be included from the June 2025 issue backwards until reaching 100 articles or until the January 2024 issue, whichever comes first. The country of the main authors (first author/last author) and the countries where all the contributors listed in the article's byline worked will be recorded. Collaboration index and degree of collaboration will be calculated. The contribution of all countries will be calculated using the Nature index's "share" concept.Depending on whether a high percentage of articles are written by authors from the same country as a given journal (and scientific society), the need to adjust the results to reflect a situation closer to reality in terms of the importance of different countries in the publication of the articles evaluated will be assessed. As a proxy, the relevance of each country in contributing to clinical pharmacology research will be calculated by multiplying the "share" score by the JCR impact factor of each journal and adding the scores obtained from the seven journals. In addition, In addition, following slightly modified terminology used by ClinicalTrials.gov, the type of sector (industry, government institutions, and 'Others') will also be recorded to help characterize the studies evaluated. However, the 'Others' category will be classified into hospitals, universities, and research centers. Funding will be recorded as public, private, and public-private.

ELIGIBILITY:
Inclusion Criteria:

* Articles on human participants, data or material. Original articles, short reports, research letters.

Exclusion Criteria:

* In vitro studies, animal studies. Editorials, letters, commentaries, perspectives.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All original research articles published in the six top clinical pharmacology hybrid journals
Sampling Method: Non-Probability Sample
Enrollment: 503 (Actual)
Dates: Start 2025-09-15 (Actual); Primary Completion 2025-11-04 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
countries where authors conducted their study | Articles of interest to be included from the June 2025 issue backwards until reaching 100 articles or until the January 2024 issue, whichever comes first
  The country of the principal authors and of all collaborators will be registered following Nature Index 'share' concept

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Dal-Re, MD, PhD, MPH, Principal Investigator — Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz
Locations (1):
- Health Research Institute Fundación Jiménez Díaz, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
All data to be used in this study are in the public domain.